CLINICAL TRIAL: NCT05696158
Title: A Prospective, Open-Label Trial of MHNA-003, a Smartphone-Delivered Cognitive Behavioral Therapy (CBT) Treatment, in Adults With Symptoms of Tinnitus
Brief Title: Mahana Tinnitus Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahana Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHNA-003-001
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2023-11

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MHNA-003 (Experimental): MHNA-003 is a self-guided digital program for people living with tinnitus
  Interventions: Device: MHNA-003

INTERVENTIONS:
Device: MHNA-003 — MHNA-003 is a self-guided digital program for people living with tinnitus
  Other Names: Mahana™ Tinnitus

SUMMARY:
The main objective of this prospective, open-label, non-significant risk study is to assess the efficacy and safety of Mahana™ Tinnitus together with care as usual in approximately 250 adults with symptoms of tinnitus.

DETAILED DESCRIPTION:
Following informed consent, all participants will complete a series of screening questionnaires to determine eligibility for study entry. Eligible participants will be enrolled, and will receive access to MHNA-003 (Mahana™ Tinnitus). Participants will use MHNA-003 for 6 weeks, completing assessments at Baseline and Weeks 2, 4, and 6 following Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Participant scores ≥ 25 on the Tinnitus Functional Index.
* Participant has experienced symptoms of tinnitus for at least 3 months.
* Participant is at least 18 years of age at the time of consent.
* Participant resides in the United States.
* Participant is able to speak, read, and understand English.
* Participant has access to an iOS or Android smartphone with the ability to complete study tasks.
* Participant is able to commit the time required to complete therapy modules and study assessments.

Exclusion Criteria:

* Participant scores ≥2 on item 9 (suicidal thoughts) of the Beck's Depression Index (BDI).
* Participant has been hospitalized for psychiatric reasons within 12 months of screening.
* Participant is currently enrolled in or plans to enroll in another clinical study that could impact outcomes of this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mahana Therapeutics, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MHNA-003
Started | 97
Completed | 57
Not Completed | 40

BASELINE CHARACTERISTICS:
Arm/Group | MHNA-003
Number analyzed (Participants) | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.84 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 85
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 97

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in TFI Score From Baseline to Week 6
Description: The Tinnitus Functional Index (TFI) is a validated, 25-item questionnaire designed to measure the severity and negative impact of tinnitus. Total scores range from 0-100 with higher scores representing higher severity and more negative impact. An improvement of 13 or more points is considered a clinically meaningful change.
Time Frame: 6 weeks
Population: Intent to treat population
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | MHNA-003
Number analyzed (Participants) | 97
score on a scale | -20.50 (1.86)

2. Primary Outcome: Tinnitus Functional Index Responder Rate
Description: The Tinnitus Functional Index (TFI) is a validated, 25-item questionnaire designed to measure the severity and negative impact of tinnitus. Total scores range from 0-100 with higher scores representing higher severity and more negative impact. A responder is defined as a participant who experienced an improvement of 13 or more points from baseline to Week 6. The responder rate is the percentage of participants considered responders at Week 6.
Time Frame: 6 weeks
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | MHNA-003
Number analyzed (Participants) | 97
percentage of responders | 61.3 [45.6 to 77.0]

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | MHNA-003
All-Cause Mortality (participants affected / at risk) | 0/97
Serious Adverse Events (participants affected / at risk) | 0/97
Other Adverse Events (participants affected / at risk) | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT05696158/Prot_SAP_000.pdf